CLINICAL TRIAL: NCT01852955
Title: Perioperative Systemic Acetaminophen to Improve Postoperative Quality of Recovery After Ambulatory Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Gildasio De Oliveira, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00078104
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Outpatient; Surgery; Breast; Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen (Active Comparator): Administration of IV acetaminophen 1000 mg over 15 minutes at the start of surgical closure.
  Interventions: Drug: IV acetaminophen
- Placebo (Placebo Comparator): Administration of placebo (sterile normal saline)group-same volume of saline solution administered in the same fashion as the acetaminophen
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV acetaminophen — Administration of IV acetaminophen 1000 mg over 15 minutes at the start of surgical closure
  Arms: IV acetaminophen
Drug: Placebo — Administration of placebo (sterile normal saline)group-same volume of saline solution administered in the same fashion as the acetaminophen
  Arms: Placebo

SUMMARY:
Recent evidence demonstrates that perioperative pain continues to be poorly managed among ambulatory surgical patients. More importantly, few interventions that minimize postoperative pain have also shown to improve patient overall quality of post-surgical recovery. Ketorolac has been used to minimize perioperative pain despite the lack of evidence for its use when administered as a single dose preventive strategy.Ketorolac has also been associated with a higher incidence of perioperative hematomas and the need for surgical re-exploration after breast surgery.

Systemic acetaminophen has become recently available in The United States. In contrast to ketorolac, systemic acetaminophen has not been reported to have adverse side effects on patients undergoing breast surgery. Although evidence suggests that a single dose perioperative acetaminophen reduces postoperative pain, it remains unknown if a single dose intravenous acetaminophen improves postoperative quality of recovery after ambulatory surgery.

The main objective of the current investigation is to evaluate the effect of a single dose systemic acetaminophen on postoperative quality of recovery after ambulatory breast surgery. We also seek to determine if systemic acetaminophen would decrease postoperative pain and the time to hospital discharge in the same population.

Significance: The current project evaluates a potential intervention to improve perioperative pain and recovery after ambulatory breast surgery. Postoperative pain in the ambulatory surgical patients has been shown consistently to be poorly managed.

DETAILED DESCRIPTION:
Patients will be recruited up to the day of surgery. They will be then randomized using a computer generated table of random numbers to two groups: Group A (IV acetaminophen 1000 mg over 15 minutes at the start of surgical closure) and Group B (placebo group-same volume of saline solution administered in the same fashion).This dose has been commonly used in other studies involving IV acetaminophen.6 Both drugs will be identical and will be prepared by hospital pharmacy. After placement of standard ASA monitors, induction will be performed with 0.1mcg/kg/min of remifentanil IV, propofol 1.5-2.5 mg/kg IV and succinylcholine 1-2 mg/kg IV. Tracheal intubation will be performed using a MAC 3 blade and a size 7 endotracheal tube. Maintenance will be achieved with remifentanil infusion titrated to keep the blood pressure within 20% of baseline values and sevoflurane titrated to keep a bispectral index monitor between 40 and 60. Patients will receive ondansetron 4mg IV and dexamethasone 4 mg IV for postoperative nausea and vomiting prophylaxis. In the recovery room patients will receive hydromorphone IV in divided doses to keep pain <4/10(scale where 0 means no pain and 10 is the worst pain) and metoclopramide 10 mg IV as rescue antiemetic. Data will be collected by a research assistant blinded to the group allocation. Data collected will involve pain at PACU arrival (NRS-0-10), presence of nausea and vomiting, severity of nausea and vomiting, total opioid consumption in PACU, time to discharge using a Modified Postanaesthetic Discharge Scoring System (MPADSS) 9, total opioid consumption 24 hours, QoR40 24hours after surgery.8

ELIGIBILITY:
Inclusion Criteria:

* Outpatient lumpectomy
* ASA I and II
* Age between 18-70

Exclusion:

* Pregnancy
* History of liver disease
* Unable to understand the informed consent
* Chronic pain with use of opioid in the last week
* Allergy to acetaminophen

Drop-out: surgeon or patient request

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gildasio De Oliveira, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] De Oliveira GS Jr, Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg. 2012 Aug;115(2):262-7. doi: 10.1213/ANE.0b013e318257a380. Epub 2012 May 14. PMID 22584558
- [Background] De Oliveira GS Jr, Ahmad S, Fitzgerald PC, Marcus RJ, Altman CS, Panjwani AS, McCarthy RJ. Dose ranging study on the effect of preoperative dexamethasone on postoperative quality of recovery and opioid consumption after ambulatory gynaecological surgery. Br J Anaesth. 2011 Sep;107(3):362-71. doi: 10.1093/bja/aer156. Epub 2011 Jun 13. PMID 21669954
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] Cawthorn TR, Phelan R, Davidson JS, Turner KE. Retrospective analysis of perioperative ketorolac and postoperative bleeding in reduction mammoplasty. Can J Anaesth. 2012 May;59(5):466-72. doi: 10.1007/s12630-012-9682-z. Epub 2012 Mar 21. PMID 22434401
- [Background] McNicol ED, Tzortzopoulou A, Cepeda MS, Francia MB, Farhat T, Schumann R. Single-dose intravenous paracetamol or propacetamol for prevention or treatment of postoperative pain: a systematic review and meta-analysis. Br J Anaesth. 2011 Jun;106(6):764-75. doi: 10.1093/bja/aer107. Epub 2011 May 9. PMID 21558067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Acetaminophen | Placebo
Started | 35 | 35
Completed | 33 | 32
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Customized [Mean (Full Range); unit: years]
  Age | 60 [54 to 65] | 52 [44 to 68] | 55 [44 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 65
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery at 24 Hours(QoR-40 Instrument)
Description: Quality of recovery score 24 hours after the surgical procedure. Total score range of 40 (poor recovery) and a score of 200 (good recovery).
Time Frame: 24 hours after the surgical procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 33 | 32
units on a scale | 189 [183 to 194] | 183 [175 to 190]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = .01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Opioid Consumption
Description: Postoperative opioid consumption over 24 hours. Converted into oral mg of morpine equivalents.
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: oral mg of morpine equivalents
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 33 | 32
oral mg of morpine equivalents | 20 [10 to 30] | 30 [10 to 40]
Statistical Analysis 1: Comparison: IV Acetaminophen vs Placebo; Test type: Superiority or Other; p = .04, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Postoperative Pain in the Post Anesthesia Care Unit
Description: Postoperative pain within the post anesthesia care unit after surgery. Area under the numeric rating scale for pain versus time curve in the post anesthesia care unit (score * min).Numeric rating scale for pain on a scale of 0-10 (0 is no pain and 10 is high pain) versus time curve in the post anesthesia care unit ( score * min). Area under a curve units of the horizontal axis multiplied by the units of the vertical axis. A higher value indicates more pain and time in the Post Anesthesia Care Unit.The range is 0 pain to x time in minutes x 1 hour to 5 hour ( 60-300 minutes) . The pain scores were collected at 15 minute intervals from the time of admission to the PACU. The area under the NRS pain scale versus time curve was calculated using the trapezoidal method as an indicator of pain burden during early recovery (Graph Pad Prism ver 5.03, Graph Pad Software INC.
Time Frame: Time in the post anesthesia care unit after surgery (average of 5 hours)
Measure: Median (Inter-Quartile Range); unit: (units on a scale * minutes
Arm/Group | IV Acetaminophen | Placebo
Number analyzed (Participants) | 33 | 32
(units on a scale * minutes | 255 [225 to 300] | 240 [180 to 300]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; p = .36, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Development of nausea 24 hours after surgery.
Arm/Group | IV Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 16/33 | 12/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen (N=33) | Placebo (N=32)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) — Vomiting within 24 hours of surgery
Nausea (Gastrointestinal disorders) | 13 (13) | 11 (11) — Nausea within 24 hours of surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No